CLINICAL TRIAL: NCT01305759
Title: Psychological, Sexually and Social Consequences of Osteoarthritis Treatment With Total Hip or Total Knee Arthroplasties and Joint Preserving Surgery
Brief Title: Psychological, Sexually and Social Consequences of Osteoarthritis Treatment With THA or TKA and Joint Preserving Surgery
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Frederiksberg University Hospital (Other); Aarhus University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Klit, MD, Hvidovre University Hospital
Other Study IDs: PhD-JK-01
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis; Depression; Hip Dysplasia
Keywords: Total knee arthroplasty; Total hip arthroplasty; Peri acetabular osteotomy; Social class; Health related quality of life
MeSH Terms: conditions — Osteoarthritis; Depression; Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- YoungTKA: Adults under 60 years who are having primary TKA
- YOUNGTHA: Adults under 60 years who are having primary THA
- PAOAarhus: Adults under 60 years who are having primary PAO

SUMMARY:
The project runs as a Ph.d. project at the Faculty of Health Sciences- University of Copenhagen.

In Denmark the investigators operate around 16.000 artificial hips and knees yearly, mainly due to osteoarthritis. The numbers has increased with 13,9% for hips and 50,7% for knees in the period 2004 to 2007. In 10% of the cases, or approximately 1.600 patients, the patient is younger than 50 years - mid-life, working, socially active and sexually active. The investigators have a tendency within in the orthopedic society to mainly focus on the technological aspects of the procedure and tend to forget that this is a key event for the patient with widespread consequences for the patient and his future life.

Hip- and knee arthroplasties is without no doubt two of the most important and successfully surgical procedures ever introduced. The economical cost for osteoarthritis treatment has exploded in the developed world over the last decade, with a yearly growth on 8%.

Because of the limited lifetime for an artificial hip or knee, this treatment can be unfortunate for the young patient. This has over the last years led to an increased interest for joint preserving surgery. Over the last twenty years it has been tried to delay the time for total hip arthroplasties for patients with hip dysplasia with the aid of Ganz osteotomy. Since this technique was introduced back in 1988, the research on the topic has had its main focus on optimizing the operation technique. So as with surgery with artificial hip or knee the investigators have a lack of knowledge regarding the social, work related, psychological and sexual aspects of this treatment.

Purpose The consequences of an artificial hip or knee joint regarding patients' social-life, work, psychological and sexual aspects gain very little attention international. The investigators apply most of our research funds exclusively to research and development of the surgical track and procedure, new prosthesis designs or coatings. The investigators find this study highly relevant because this kind of studies has been preformed for several chronic diseases but not osteoarthritis and its treatment.

With this study the investigators wish to examine the social, work related, psychological and sexual aspects of end stage osteoarthritis. This will lead the way for improved information to the patient and improve the surgeons' possibilities for chosen the correct time for surgery.

DETAILED DESCRIPTION:
In Denmark approximately 16.000 artificial hips or knees are inserted yearly. A increasing number that probably will continue to increase due to demographic factors and the populations rising demands on a active life in the old age. However of the 16.000 artificial joints approximately 10% are inserted in patients under fifty years(1;2). This group of patients is mid-life and thereby for most parts working and socially- and sexually active.

Total hip arthroplasty(THA) or total knee arthroplasty(TKA) is unquestionably one of the most successfully operations there has been introduced, and is capable of relieving pain, optimizing the function of the joint and optimizing the quality of life(3;4). In the resent years the main focus has been on optimizing the surgical track, whereby most of the patient today are only admitted to the hospital in 1-2 days. This progress has had a tremendous impact on patients, the departments and the health care system. Joint replacement surgery with THA or TKA is a key event for the patient and can recreate the patient's mobility but as well has widespread (but still undocumented) consequences for the patient and his future life.

In the preoperative treatment and planning of the correct time of surgery, it is imported to know, how the patient is affected of a disabling joint disease like end-stage osteoarthritis(OA) and which consequences it has to the patient to have an artificial joint. It is known, that patients with OA has a two-fold increased risk of depression(8-13).

These aspects of the treatment has so far not had the desirable attention, neither national or international At Hvidovre Hospital, Frederiksberg Hospital and Køge Hospital the Orthopaedic departments has many years of experience with joint replacement surgery at specialist level. The structures of the departments are based on modern fast-track principals, with clearly defined goals for preoperative information, pre- and postoperative regimes and discharged criteria. Thereby insuring a smooth course, short rekonvalens and a minimizing of complications.

Because of the limited lifetime for an artificial hip or knee, this treatment can be unfortunate for the young patient. This has over the last years led to an increased interest for joint preserving surgery. Over the last twenty years it has been tried to delay the time for total hip arthroplasties for patients with hip dysplasia with the aid of Peri Acetabular Osteotomy(PAO). Hip dysplasia is seen equally in both sexes. However it is more often symptomatic in females(14). In Denmark PAO is performed at Copenhagen University Hospital, Odense University Hospital and Aarhus University Hospital. The procedure is preformed on symptomatic (mainly sharp groin pain) patients in hope of delaying the development of OA. Femoroacetabular impingement (FAI) is believed to be the pathology, where repeated trauma to the acetabular labrum and adjacent chondral structures can result in labral tears and chondral delamination, leading to groin pain and over time OA. However there are only a few minor studies concerning which impact this procedure has on the young patients life in term of psychological, sexually and social wellbeing.

Patients included are both men and women from twenty to sixty years old who are admitted to undergo primary uni- or bilateral THA or TKA at Hvidovre Hospital, Frederiksberg Hospital or Køge Hospital as a result of end-stage OA, rheumatoid arthritis or another joint disease diagnosed by one of the departments doctors with specialty in joint replacement surgery. The included patients in the PAO study has all had PAO at Aarhus University Hospital between 1999-2002 and were at the age of fifteen or more at the time of surgery. To avoid co-morbidity confounders the joint disease has to be the only main disease.

The goal of the study is to investigate:

1. What are the Health-Related-Quality-Of-Life(HRQoL) consequences of end-stage hip or knee OA? The investigators will examine this with SF-36, a standardized and validated questionnaire that explores HRQOL.
2. What is the relation between the pre- and postoperative joint function and the patients HRQoL, and do this relation reflects the patient's social class and attachment to the workforce.
3. Which preoperative parameters have the strongest relation on the postoperative out-come? The highly nuanced picture the investigators get of the patients pre- and postoperative condition will enable us to answer this question.
4. How is the patient's relation to the workforce-affected by the patient's joint disease and operation? Are the investigators able to operate the patient back in work? Do the patient lose he's job because of the operation? Do the patient's with a job preoperative keep their job will those without a job preoperative do not recover their working ability because of the operation?
5. It is known that patients with OA has a two fold increased risk of depression. Is the depression due to the patients underlying disease? Or is the depression due to modulations in pain perception which lead to a lower pain threshold that again leads to the increased prevalence of symptomatic OA? If the THA or TKA is curative for the patient's depression, the investigators may assume that the depression is due to the patients disabling disease and vice versa.
6. It is known that patients with hip OA experience sexual-problems. How is this affected by joint replacement surgery? A Danish study has shown that older men -average age 70 years- who receives a THA has a highly increased risk of postoperative impotence -26% compared to the expected 3% for an age matched group. Other studies have shown that females experience an improvement of there sexual-life after THA. Unfortunately, there are only quite few and small studies concerning these subjects. The investigators wish to explore these subjects and the similar subjects for TKA, this has not previously been explored.
7. Over the last three decades there has been an increasing focus on joint preserving surgery, mainly in the form of PAO. This procedure is preformed on public hospitals in Aarhus University Hospital, Odense University Hospital and Copenhagen University Hospital. Aarhus University Hospital holds the leading experience in Denmark and performs approximately 75 procedures a year. However there is now documentation on how this procedure affects the patients HRQoL or sexual-life.

The main part of this study runs as a prospective questionnaire based study of the patients, which are having a THA or TKA at Hvidovre University Hospital, Frederiksberg University Hospital and Køge Hospital. A smaller part of the study is a retrospective questionnaire based study of the patients, which in the period 1999-2002 underwent PAO at Aarhus University Prior to planned surgery with THA or TKA the patient receive a questionnaire. This will be followed by a questionnaire 3, 6 and 12 months postoperative. Twelve months postoperative the patient will have and ambulatory control.

The patients who underwent PAO at Aarhus University Hospital in the period 1999-2002 are posted a questionnaire.

The inclusions of patients started April 2010 and runs at least to the summer of 2011 or when at least 250 patients are included.

The results are expected to be published in international English language journals and the research and findings will be defended as a PhD ad the Faculty of Health Sciences- University of Copenhagen.

Purposes of the study:

Primary purpose:

To investigate how end-stage OA and joint replacement surgery affects the patients HRQoL and herby which impact this procedure has on the young patients life in term of psychological, sexually and social wellbeing. Next the investigators wish to investigate how the patients' attachment to the workforce is affected bye end-stage OA and joint replacement surgery

Secondary purpose:

To investigate how patients with other disabling joint diseases with need for joint replacement surgery is affected as described above.

Tertiary purpose:

Edification of a database to reveal complications over years for this well-defined young patient population, who has a higher demand to there prosthesis and as a consequence put them to a higher stress.

Other purposes:

To investigate which impact PAO has on the young patients life in term of HRQoL, psychological, sexually and social wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Patients born from 01.01.1950, who are submitted fore primary THA or TKA on Hvidovre University Hospital, Frederiksberg University Hospital or Køge Hospital.
* The patient has to be capable of understanding Danish
* The patient has to be mental well an capable of understanding the information
* The patient must not have other major diseases

Exclusion Criteria:

* Terminal diseases
* Lack of ability to follow the department's standard procedures

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young adults undergoing TKA/THA/PAO with now other major health complications.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
SF-36 | 3 years
  1. What are the Health-Related-Quality-Of-Life(HRQoL) consequences of end-stage hip or knee OA? We will investigate this with SF-36, a standardized and validated questionnaire that explores HRQOL

SECONDARY OUTCOMES:
social class | 3 years
  2. What is the relation between the pre- and postoperative joint function and the patients HRQoL, and do this relation reflects the patient's social class and attachment to the workforce.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Klit, Dr, Study Director — Hvidovre University Hospital, Copenhagen, Denmark
Locations (1):
- Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark